CLINICAL TRIAL: NCT02366741
Title: Neurocognitive Function Changes in Patients With LD Small Cell Lung Cancer Undergoing Prophylactic Whole Brain Radiotherapy With Hippocampal Sparing - a Pilot Study
Brief Title: Neurocognitive Function After Prophylactic Cranial Irradiation & Hippocampal Sparing in LD SCLC Patients - a Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Leor Zach, MD, Director of the Neuro-Oncology service, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SMC-1476-14
Record Dates: First submitted 2015-01-29; First posted 2015-02-19 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Carcinoma, Small Cell
Keywords: SCLC; Neuro-cognitive function; PCI; Hippocampal sparing
MeSH Terms: conditions — Carcinoma, Small Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pilot group (Other): Five eligible patients will undergo WBRT with reduced dose to the hippocampi and will be evaluated prospectively by neuro cognitive testing, MRI scans and blood tests.
  Interventions: Radiation: Whole brain radiotherapy with reduced dose to the hippocampi

INTERVENTIONS:
Radiation: Whole brain radiotherapy with reduced dose to the hippocampi — VMAT plan to treat the whole brain while reducing the dose to the hippocampi.

SUMMARY:
Small cell lung cancer (SCLC) harbors a high risk for brain metastases. Prophylactic whole brain radiotherapy (PCI)) is the standard treatment for these patients after completing chemo-radiotherapy to the chest, with a 5% survival advantage. Recent data suggest minimal risk for hippocampal involvement in these patients. There is no published data thus far testing the effect of hippocampal sparing during WBRT on the patient's neuro-cognitive function, QOL, and survival.., The goals of the proposed study are to assess prospectively the neurocognitive changes in patients with LD SCLC who are candidates for PCI before, and periodically after PCI

DETAILED DESCRIPTION:
Background and rational Prophylactic cranial irradiation Small cell lung cancer (SCLC) is an aggressive type of lung cancer, with high sensitivity to chemotherapy and radiotherapy but with high incidence of local and distant recurrences. The brain is a common site of metastases from SCLC with a risk of up to 70% for brain involvement [1]. Prophylactic cranial irradiation (PCI) is the standard treatment for patients with limited disease (LD) SCLC after completing chemo-radiotherapy to the chest. The treatment includes whole brain radiotherapy (WBRT), reduces the incidence of brain metastases and improves overall survival (OS) by 5% [1]. The down side of WBRT is that the central nervous system (CNS) is vulnerable to radiotherapy (RT) and its related toxicity may be associated with irreversible cognitive dysfunction [2].

Radiotherapy and neuro-cognitive function It has been demonstrated that there are two main regions of human containing multipotent neural stem cells (NSCs): the subgranular zone (SGZ) within the dentate gyrus of the hippocampus, and the subventricular zone (SVZ) on the lateral aspect of the lateral ventricles [3,4,5,6,7,8]. These NSCs are capable of replacing adult neuron loss caused by various forms of harm (e.g. local ischemia, brain trauma, and radiation exposure and neurodegenerative diseases). However, they are extremely sensitive to X-rays, and thus reduction of NSCs may play an important role in radiation-induced neurocognitive impairment [6,7,8]. Neurocognitive function (NCF) has a major impact on QOL and has been actively studied in brain tumor patients treated with radiotherapy. Many studies have evaluated the neurocognitive outcome of patients treated with radiation for brain metastases and primary brain tumors [9,10,11,12,13,14]. Radiation primarily causes coagulation necrosis of the white matter tracts and cerebral vasculature by axonal demyelination and damage to vascular endothelial cells. Radiation has been shown to negatively affect various neuropsychological domains. WBRT has been shown to have greater neuropsychological impairment than focused radiation treatment [14]. Correlation, between radiation dosage to the bilateral hippocampi and impairment of NCF, was found in adult patients with benign or low-grade brain tumors treated with fractionated stereotactic radiotherapy (FSRT) [14].

An ongoing clinical trial of the radiation oncology group (RTOG) is testing the applicability of hippocampal sparing and its impact on neurocognitive changes in cancer patients with brain metastases.

Neuro-cognitive function testing Even though many studies have evaluated NCF in relation to radiation, there is no consensus regarding standardization of tests selection, time points for evaluation and correlations with biomarkers. Many studies use the Folstein Mini-Mental State Examination (MMSE) to assess neurocognitive function [15,16]. The MMSE is not a sensitive tool for detecting cognitive impairment and does not measure the cognitive functions affected by radiation. The NeuroTrax system is described elsewhere [17]. In brief, Mindstreams consists of custom software that resides on the local testing computer and serves as a platform for interactive cognitive tests that produce accuracy and reaction time (millisecond time-scale) data. In case of conducting several trails for a single patient, Mindstreams uses a different version of the tests in each trial, in order to avoid a learning bias. Tests are available in multiple languages, and equivalence among English and Hebrew versions has been shown [17]. After tests are run on the local computer, data are automatically uploaded to a central server, where calculation of outcome parameters from raw single-trial data and report generation occurs. All responses are made with the mouse or with the number pad on the keyboard. Participants are familiarized with these input devices at the beginning of the battery, and practice sessions prior to the individual tests instruct them regarding the particular responses required for each test.

Hippocampal sparing during PCI Recent data suggest minimal risk for hippocampal involvement in patients with SCLC and brain metastases suggesting that reduced radiation dose to these areas during PCI would not significantly compromise the control in the brain [18]. There is no published data thus far testing the effect of hippocampal sparing during PCI on the patient's neuro-cognitive function, QOL, and survival. Volumetric arc radiotherapy (VMAT) and intensity modulated radiotherapy (IMRT) use advanced radiation planning software with computerized algorithms of inverse planning to allow differential radiation dose distribution within the same radiation field. A preliminary dosimetric work in the radiation oncology unit at Sheba medical center has proved the feasibility of generating WBRT plans using these techniques while reducing the dose to the hippocampi. The investigators compared 3 radiotherapy plans (standard 2 lateral field plan, IMRT plan and a VMAT plan) aiming to give 30Gy to the brain, with 40Gy integrated boost to evident brain metastases (using magnetic resonance imaging - MRI scan) and reduced dose to the hippocampi (<10Gy) according to RTOG 0933 protocol. IMRT achieved better results in general then the VMAT plans, especially in patients with brain metastases located closer to the hippocampi. The work has been presented in the EANS European Association of Neuro-Surgeonsmeeting last year.

Serum biomarkers for CNS damage Neuron-specific enolase (NSE) and S100 are two serum tumor markers that may be used as a potential screening tool for brain injury caused by radiation [19-27]. NSE is a glycolytic enzyme found in the CNS, expressed by neural and neuroendocrine cells. Elevated levels of NSE have been found in patients with brain metastases from NSCLC. A multi-center retrospective study involving 231 NSCLC patients demonstrated that high serum levels of NSE indicated shorter survival and was a specific marker of metastases. It is thought that the rise in NSE in brain metastasis patients reflects the extent of neuronal damage, as seen following a cerebral stroke. S100 protein is a nervous-system-specific cytoplasmic protein found in astrocytes and released into the serum when the blood brain barrier (BBB) is breached. Brain metastases were shown to be associated with elevated levels of S100 in several malignancies. Serum S-100B has also been demonstrated to be useful in determining brain damage related to stroke.

Imaging biomarkers for CNS damage Although brain radiotherapy induces white matter changes which can be depicted in standard MRI scans, no correlation was found between these changes and cognitive impairment. BBB disruption is an early, readily recognizable pathophysiological event occurring after radiation injury. It is detectable in vivo/in vitro by MRI and other imaging modalities, and appears to precede white matter necrosis. Micro-vascular leakage (MVL), calculated from perfusion MRI, is more sensitive than conventional contrast-enhanced MRI to subtle BBB opening, reflecting abnormal permeability of immature vessels. Treatment response assessment maps (TRAM) is a novel methodology, based on T1-MRI acquired up to 90 min after contrast injection, which allows depiction of subtle BBB disruption [28]. The resulting calculated maps, depict BBB functioning of the full brain, with high spatial resolution and high sensitivity to subtle BBB abnormalities. Results in >200 patients with primary and metastatic brain tumors demonstrate the high sensitivity for subtle BBB disruption and the ability of the investigators maps to depict and differentiate various BBB disruption patterns within the tumor and the irradiated area.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with histologically confirmed LD SCLC and complete response (CR) of the primary lesion after chemo-radiotherapy to the chest and who are candidates for PCI will be accrued

Exclusion Criteria:

* A history of malignant disease other then SCLC
* Previous cranial irradiation
* Medical or social condition which limits the ability of the patient to undergo neuro-cognitive testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients that complete a year of imaging, neuro-cognitive and clinical follow up after WBRT with HC sparing as a measure of feasibility to conduct a randomized study in this patient population. | 1 year

SECONDARY OUTCOMES:
Number of patients with no changes in the neurocognitive tests score and QOL as a measure for the correlation between NCT and HC sparing. | 1 year
Number of patients with no changes in serum markers for neuronal damage and as a measure for reduced damage due to hippocampal sparing | 1 year
Number of patients with changes in imaging biomarkers (TRAM) and neurocognitive tests score decline as a measure for a potential correlation between the two. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Leor Zach, MD, Principal Investigator — Director of the Neuro-Oncology service
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel